CLINICAL TRIAL: NCT00290862
Title: A Randomized, Controlled Clinical Study to Evaluate the Safety and Effectiveness of CORTOSS® Synthetic Cortical Bone Void Filler in Vertebral Augmentation
Brief Title: A Safety and Efficacy Study for Treatment of Painful Vertebral Compression Fractures Caused by Osteoporosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Orthovita d/b/a Stryker (Industry)
Responsible Party: Maarten Persenaire, M.D., Chief Medical Officer, Orthovita
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1100-0008
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Spinal Fractures
Keywords: Osteoporosis; Spine fracture; Back Pain; Vertebroplasty; Vertebral compression fractures related to osteoporosis
MeSH Terms: conditions — Spinal Fractures; Osteoporosis; Back Pain

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- CORTOSS (Experimental): Patients prospectively randomized to be treated with Cortoss constitute treatment group.
  Interventions: Device: Percutaneous Vertebral Augmentation of compression fractures
- PMMA (Active Comparator): Patients prospectively randomized to be treated with PMMA constitute active control group.
  Interventions: Device: Percutaneous Vertebral Augmentation of compression fractures

INTERVENTIONS:
Device: Percutaneous Vertebral Augmentation of compression fractures — Study eligible patients with painful osteoporotic compression fractures will be randomized to percutaneous vertebroplasty with CORTOSS (treatment group) or PMMA (active control group).
  Other Names: CORTOSS, a Bis-GMA composite material, a vertebral augmentation strengthening agent.; PMMA, commercially available poly methyl methacrylate material, on-label for vertebral augmentation.

SUMMARY:
Doctors are studying an investigational treatment to be used during the vertebroplasty procedure when treating vertebral compression fractures (spine fractures) that may help to reduce pain and restore mobility. If one has experienced back pain for at least 4 weeks but not longer than 1 year, he/she may be eligible to participate.

The purpose of this protocol is to describe the methods for the clinical evaluation of Cortoss for vertebroplasty in patients with painful osteoporotic compression fractures.

Eligible patients with painful osteoporotic compression fractures of the spine are divided into two groups. Each enrolled patient will have the vertebroplasty procedure; however one group of patients will have the vertebroplasty procedure using polymethylmethacrylate [PMMA] (a Food and Drug Administration [FDA]-approved bone cement) and the other group of patients will have the vertebroplasty procedure using a relatively new (investigational) biomaterial called Cortoss.

DETAILED DESCRIPTION:
This is a prospective, multi-center randomized, controlled study designed to evaluate the safety and effectiveness of Cortoss® Synthetic Cortical Bone Void Filler in vertebral augmentation using the percutaneous vertebroplasty technique. Study eligible patients with painful osteoporotic compression fractures will be randomized (2:1) to vertebroplasty with Cortoss (treatment group) or PMMA (control group), respectively. Patients will not be told which treatment they will receive (single blind study design). Safety and effectiveness will be determined by comparing the success rate of the treatment group to the success rate of the control group. Secondary endpoints will include Quality of Life, Patient satisfaction, evaluation of the patient's pain and function post-operatively compared to baseline, and maintenance of vertebral body height and alignment.

For the purposes of this study, vertebral augmentation, or vertebroplasty, is defined as a minimally invasive procedure utilizing manual instruments and radiological guidance to deliver an in-situ polymerizable material to stabilize a collapsed or fractured vertebral body. The goal is to alleviate pain caused by the fracture and enhance or prevent further deterioration of function.

This multi-center study will evaluate Cortoss for the augmentation of one or two vertebra(e), fractured as a result of osteoporosis, located between (and including) the levels of the sixth thoracic and the fifth lumbar vertebrae. A total of 243 patients will be enrolled at up to 19 sites. All subjects must have radiographic evidence of a vertebral body fracture due to osteoporosis. After complying with all eligibility criteria, subjects will sign an informed consent document and will be randomized into vertebroplasty treatment with Cortoss or PMMA (1:1 ratio). Patients will be followed for at least 24 months and recruitment is expected to take between 9 and 12 months. Visits and assessments are planned according to the time and events schedule.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age
* Have sustained a painful osteoporotic vertebral compression fracture (VCF) for at least 4 weeks but no longer than 1 year or have radiographic evidence of at least 5% worsening vertebral collapse as compared to previous radiographic evidence
* Give written Informed Consent to participate in the study and be willing to comply with protocol requirements
* Have pain requiring the regular use of analgesics or have a substantially altered life-style due to pain or disability
* Have central pain over the spinous process upon palpation at the planned level(s)
* Are appropriately communicative to verbalize and differentiate with regard to location and intensity of their pain
* Are physically and mentally willing and able to comply with the clinical and radiographic follow-up schedule
* Have radiographic evidence of one or two, Grade 1 or greater according to Genant's criteria, osteoporotic VCF(s) between (and including) the level of the sixth (6th) thoracic to the fifth (5th) lumbar
* Have an acute or persistent (not healed) fracture demonstrated by magnetic resonance imaging (MRI) or bone scan
* Have a patient self-assessment VAS score >= 50 mm at the pre-treatment visit
* Have a 30% or greater disability score on the baseline ODI (version 2.0).

Exclusion Criteria:

* Have significant vertebral collapse defined as more than 70% of original vertebral height, or a burst or pedicle fracture with posterior cortical wall disruption
* Have posterior vertebral wall displacement occupying more than 20% of the cross sectional area of the spinal canal
* Have neurologic symptoms or deficits, or radiculopathy related to the VCF
* Have pain based on a clinical diagnosis of herniated nucleus pulposus, high energy trauma, severe spinal stenosis as evidenced by progressive weakness or paralysis, or bone tumor at the level(s) of pathology as evidenced by computed tomography (CT) scan
* Have indications of instability related to the VCF at the level to be treated (e.g., neurologic deficit, kyphosis > 30º, translation > 4 mm, and/or interspinous process widening)
* Have canal compromise causing clinical manifestations of cord, neural foramen, or nerve root compression at the level(s) to be treated
* Have a bleeding disorder, including coagulopathy
* Have severe cardiopulmonary deficiencies
* Have an active systemic or local infection
* Are currently being treated for cancer or HIV
* Have a known allergy to acrylics (e.g., methyl methacrylate)
* Subject is currently an alcohol, solvent or drug abuser
* Female patients who are pregnant or nursing, or of childbearing potential not using a reliable contraceptive method
* Are involved in medical litigation
* Are prisoners
* Have participated in another investigational study within 30 days prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2004-09; Study Completion 2009-03

PRIMARY OUTCOMES:
Early and sustained decrease in pain (efficacy prong of primary endpoint) at 24 months compared to pre-treatment baseline using the Visual Analog Scale (VAS) | 24 Months
Maintenance or improvement in function (efficacy prong of primary endpoint) at 24 months compared to pre-treatment baseline using the Oswestry Disability Index (ODI) | 24 Months
Maintenance vertebral height and alignment (efficacy prong of primary endpoint) at 24 Months compared to 1-month post-vertebropalsty baseline radiographs | 24 Months
No device-related subsequent surgical intervention at study treated level | 24 Months

SECONDARY OUTCOMES:
Maintenance or improvement in quality of life (secondary endpoint) at 24 months compared to baseline using the SF-12 | 24 Months
Ambulatory status | 24 Months
Patient satisfaction | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Persenaire, M.D., Study Director — Orthovita, Inc.
Locations (18):
- United States (18):
  - Scottsdale Medical Center, Scottsdale, Arizona
  - Core Orthopaedic Medical Center, P.C., Encinitas, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - St. John's Spine Institute, Santa Monica, California
  - Indian River Radiology, Vero Beach, Florida
  - Emory Orthopaedics and Spine Center, Atlanta, Georgia
  - Millenium Pain Center, Bloomington, Illinois
  - Northwestern University, Chicago, Illinois
  - The Spine Institute of Louisiana, Shreveport, Louisiana
  - Washington University Medical Center, St Louis, Missouri
  - Hospital for Special Surgery (HSS), New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Mission Hospitals, Asheville, North Carolina
  - Dayton Interventional Radiology, Kettering, Ohio
  - Edmond Medical Center, Oklahoma City, Oklahoma
  - Mercy Health Center, Oklahoma City, Oklahoma
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Endovascular Center of Houston, Houston, Texas